CLINICAL TRIAL: NCT01079598
Title: A Prospective Multicenter Study on the Treatment of Incompetent Perforators With the VNUS® Closure Radiofrequency Stylet
Brief Title: RFS (Radiofrequency Stylet) - Radiofrequency Perforator Vein Treatment Study
Acronym: TRIPLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFS-09-01
Record Dates: First submitted 2010-02-24; First posted 2010-03-03 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Venous Insufficiency
Keywords: IPV; RadioFrequency; QOL
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): RF ablation with ClosureRFS Stylet
  Interventions: Device: RF Ablation (ClosureRFS Stylet)

INTERVENTIONS:
Device: RF Ablation (ClosureRFS Stylet) — Bipolar energy radiofrequency ablation with RFS stylet
  Other Names: RFS; RFS Stylet; ClosureRFS Stylet

SUMMARY:
The purpose of this study is to demonstrate that patients will improve the immediate treatment outcomes from successive radiofrequency ablation (RFA) of incompetent perforator veins (IPVs).

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that patients who have competent great saphenous vein (GSV) and short saphenous vein (SSV) or have undergone prior successful endovenous treatment of an incompetent GSV and/or SSV but continue to demonstrate clinical symptoms of peripheral venous insufficiency resulting from incompetent perforator veins (IPVs) will improve the immediate treatment outcomes from successive radiofrequency ablation (RFA) of IPVs veins.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18 to 80 years, from all racial and ethnic origin
* Have the ability to understand the requirements of the study, provide written informed consent to participate, and agree to abide by the study requirements
* Available for all the follow-up visits and in a physical condition allowing ambulation after the procedure
* Incompetent GSV and/or SSV in the target limb has been treated at least 3 months before study enrollment or competent GSV and SSV at time of treatment
* CEAP 4 - 6 classification
* DUS reflux of ≥0.35 sec or more of the target IPV and/or an intra-fascia diameter of ≥0.3 mm

Exclusion Criteria:

* Acute (at Screening) superficial venous thrombosis of either limb
* Acute (within the prior 3 months) deep venous thrombosis or phlebitis in either limb
* Complete or near complete deep venous obstruction documented by ultrasound
* Previously participated in any study involving ClosureRFS
* Actively participated in any other investigational study within 30 days of enrollment into this study
* Pregnant at the time of treatment. Status verified by pregnancy test via blood or urine for women ≤ 55 years old.
* Having a medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all required study follow-up
* Have any condition that, in the opinion of the Investigator, would jeopardize the safety of the patient or affect the validity of the trial results
* Have a history of excessive alcohol consumption or any use of illegal drugs rendering the patient unreliable, or at risk during this trial
* Have undergone major surgery which may result in abnormalities of the target body area, reasonably suspected to compromise the study outcomes
* Have undergone an invasive procedure of the target body area (e.g., needle biopsy or surgical procedure) within 30 days of enrollment into this study
* Known incompatibility, such as an allergic reaction to anesthetics to be used in the incompetent perforator vein treatment
* Patients requiring hyperbaric therapy involving the treated limb during the 6 month post treatment follow-up period
* Great toe pressure measurement of ≤ 70 mmHg
* CEAP 6 classified patients receiving high dose steroid medication or the following medications that interfere with normal mechanisms of wound healing, e.g. glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), anti-neoplastic and immunosuppressive drugs, and others like, colchicine and penicillamine.
* Expressing a body mass index (BMI) of ≥ 35.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hasenbank, PhD, Study Director — Medtronic
Locations (3):
- United States (3):
  - Varicosity Vein Center, Birmingham, Alabama
  - Vein Care Pavilion of the South, Evans, Georgia
  - Allegiance Vascular Health, Jackson, Michigan

IPD SHARING:
Plan to Share IPD: No
Out of a planned 225 patient subject size, a total of 8 subjects were enrolled with 10 limbs treated. As a result of stagnant enrollment in the study, a decision was made to terminate the study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: RF ablation of incompetent perforator and tributary veins with ClosureRFS Stylet
Period: Overall Study
Arm/Group | Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life and Clinical Assessments Compared to Pretreatment Baseline.
Description: QOL and clinical assessments measured by periodic CIVIQ2 and VCSS assessments were planned to be compared at each follow-up visit to pretreatment baseline. However, with the very low enrollment and limited data available, analysis and study results are inconclusive.
Time Frame: 6 months
Population: Analysis was not able to be completed due to very low enrollment and limited data available. No results available.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Cessation of Flow Through the Perforator Vein
Description: Cessation of incompetent flow and reflux is defined as the absence of blood flow within the treated segment of the perforator vessel at the level the vessel crosses the superficial fascia. Key measures that will be used to evaluate the intervention that are a focus of the study.
Time Frame: 6 months
Population: Analysis was not able to be completed due to very low enrollment and limited data available. No results available.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: CEAP Classification (Clinical Severity, Etiology or Cause, Anatomy, Pathophysiology)
Description: CEAP Classification at Month 6 will be reported.
Time Frame: 6 months
Population: Analysis was not able to be completed due to very low enrollment and limited data available. No results available.
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Cessation of Flow Reflux Through the Perforator Vein
Description: as for outcome 2
Time Frame: 6 months
Population: Analysis was not able to be completed due to very low enrollment and limited data available. No results available.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Enrollment through study completion
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Thrombus Extension (Vascular disorders) | 1 (1) — One subject developed a thrombus extension into the tibial vein post perforator ablation that was discovered during the 3-day follow-up visit by DUS exam. The patient was placed on anti-platelet medication and the outcome was reported as resolved.

LIMITATIONS AND CAVEATS:
Limitations of the study, such as early termination leading to small numbers of participants analyzed and technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less